CLINICAL TRIAL: NCT05177588
Title: Efficacy of Metformin as add-on Therapy in Non-Diabetic Heart Failure Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Sayed Kamel, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL (2582)
Record Dates: First submitted 2021-12-16; First posted 2022-01-04 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
Keywords: Metformin; Heart failure; Non-diabetic; left ventricular mass index
MeSH Terms: conditions — Heart Failure | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: This is a prospective, interventional, randomized controlled, open label study. The study sample will include heart failure patients with pre-diabetes
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Patients in the metformin group will receive a starting dose of 1000 mg/day. The dose will be titrated as tolerated to a maximum of 2000 mg/. Patients will receive the medications for six year and will be followed up for the duration of the study. Patients will be assessed at baseline, 3 months, and 6 months.
  Interventions: Drug: Metformin Hydrochloride
- Standard of Care (No Intervention): Patients in the control arm will continue the SOC medications

INTERVENTIONS:
Drug: Metformin Hydrochloride — Metformin 2000 mg/day
  Other Names: Glucophage; Cidophage
  Arms: Metformin

SUMMARY:
There is an increasing interest in the use of metformin in CV diseases and there is an increasing interest in studying its potential new roles in heart failure patients. There were some concerns related to the safety of metformin in such diabetic patients due to the risk of lactic acidosis. However, recent studies showed that metformin was safe or even beneficial in HF patients. We hypothesized that metformin might improve morbidity, mortality, cardiac function, and HR-QoL in non-diabetic patients with HFrEF.

DETAILED DESCRIPTION:
Metformin is an anti-diabetic drug that is known improve insulin sensitivity and reduce insulin resistance. A published meta-analysis of randomized controlled trials (RCTs) reported a reduction of weight and insulin resistance in metformin users. Animal models also showed that metformin reduces cardiac hypertrophy. Observational studies showed a beneficial effect for metformin in patients with type 2 diabetes mellitus (T2DM) and heart failure. A recent study found that metformin reduced oxidative stress in non-diabetic patients with CAD.

Metformin has multiple modes of actions involving both AMP-activated protein kinase (AMPK) dependent and AMPK-independent mechanisms that may be implicated in cardiac hypertrophy. At the systemic level, a review of clinical and experimental data showed that metformin improves endothelial function, protects from oxidative stress and inflammation, as well as the negative effects of angiotensin II. Observational studies also reported cardiovascular benefits in metformin users especially in patients with type 2 diabetes mellitus (T2DM) and heart failure. Metformin has also been shown to exert a cardio protective effect and it has been shown to reduce oxidative stress which is a common finding in heart failure patients. For these reasons, there is an increasing interest in the use of metformin in CV diseases and there is an increasing interest in studying its potential new roles in this aspect. We hypothesized that metformin might improve morbidity, mortality, cardiac function, and HR-QoL in non-diabetic patients with HFrEF.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure (>6 months duration)
* Stabilized on recommended or maximally tolerated dose of ACE-I/ARB or ARNI (unless contraindicated) and beta-blocker (unless contraindicated). If indicated, an aldosterone receptor antagonist should be given (unless contraindicated).
* Reduced ejection fraction defined as LVEF < 45%
* NYHA-class II or III or IV with stable symptoms for at least the past 3 months
* Creatinine clearance > 45 ml/min

Exclusion Criteria:

* Diabetes mellitus: Diabetes will be diagnosed using the 2018 The American Diabetes Association (ADA) "Standards of Medical Care in Diabetes 15

  * FPG ≥126 mg/dL (7.0 mmol/L). Fasting is defined as no caloric intake for at least 8 h.*
  * 2-h PG ≥200 mg/dL (11.1 mmol/L) during OGTT. The test should be performed as described by the WHO, using a glucose load containing the equivalent of 75-g anhydrous glucose dissolved in water.
  * A1C ≥6.5% (48 mmol/mol). The test should be performed in a laboratory using a method that is NGSP certified and standardized to the DCCT assay.*
  * In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥200 mg/dL (11.1 mmol/L).
* Any oral or injectable hypoglycemic therapy (e.g. insulin, sulfonylureas)
* Recent Hospitalizations in the past 3 months
* Metformin treatment within the last 3 months
* Creatinine clearance below 45 in the prior 6 months as assessed by Cockcroft and Gault equation
* Known allergy to metformin or major side effects to metformin treatment
* Atrial fibrillation with poorly controlled ventricular rate at rest (> 100 beats/min)
* Hypertrophic cardiomyopathy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in total antioxidant capacity (relative and absolute) | 6 months
  Change Total antioxidant capacity as assessed by colorimetric assay
Change in Malondialdehyde (MDA) | 6 months
  Change in Malondialdehyde (MDA) as assessed by colorimetric assay
Chagne in left ventricular mass index | 6 months
  Chagne in left ventricular mass index as assessed by Echocardiography

SECONDARY OUTCOMES:
Chagne in Ejection Fraction | 6 months
  Ejection fraction as assessed by echocardiography
New York Heart Association functional classification (NYHA): | 6 months
  The NYHA classifies patients in one of four possible categories based on the physical activity limitations; the limitations/symptoms are in regards to normal breathing andvarying degrees in shortness of breath and or angina pain
TAC | 6 months
  Total antioxidant capacity as assessed by colorimetric assay
MDA | 6 months
  MDA as assessed by colorimetric assay
Adverse reactions of metformin | 6 months
  Incidence of lactic acidosis
Change in fasting blood glucose (FBG) | 6 months
  Change in FBG from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Kamel, MSc., Principal Investigator — Faculty of Pharmacy, Cairo University
Locations (1):
- Agouza Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larsen AH, Jessen N, Norrelund H, Tolbod LP, Harms HJ, Feddersen S, Nielsen F, Brosen K, Hansson NH, Frokiaer J, Poulsen SH, Sorensen J, Wiggers H. A randomised, double-blind, placebo-controlled trial of metformin on myocardial efficiency in insulin-resistant chronic heart failure patients without diabetes. Eur J Heart Fail. 2020 Sep;22(9):1628-1637. doi: 10.1002/ejhf.1656. Epub 2019 Dec 21. PMID 31863557
- [Background] Mohan M, Al-Talabany S, McKinnie A, Mordi IR, Singh JSS, Gandy SJ, Baig F, Hussain MS, Bhalraam U, Khan F, Choy AM, Matthew S, Houston JG, Struthers AD, George J, Lang CC. A randomized controlled trial of metformin on left ventricular hypertrophy in patients with coronary artery disease without diabetes: the MET-REMODEL trial. Eur Heart J. 2019 Nov 1;40(41):3409-3417. doi: 10.1093/eurheartj/ehz203. PMID 30993313
- [Derived] Kamel AM, Ismail B, Abdel Hafiz G, Sabry N, Farid S. Effect of Metformin on Oxidative Stress and Left Ventricular Geometry in Nondiabetic Heart Failure Patients: A Randomized Controlled Trial. Metab Syndr Relat Disord. 2024 Feb;22(1):49-58. doi: 10.1089/met.2023.0164. Epub 2023 Oct 10. PMID 37816240
- [Derived] Kamel AM, Ismail B, Abdel Hafiz G, Sabry N, Farid S. Total Antioxidant Capacity and Prediabetes Are Associated with Left Ventricular Geometry in Heart-Failure Patients with Reduced Ejection Fraction: A Cross-Sectional Study. Metab Syndr Relat Disord. 2023 Jun;21(5):282-291. doi: 10.1089/met.2023.0019. Epub 2023 May 23. PMID 37220008